CLINICAL TRIAL: NCT03662386
Title: Prospective Analysis of "Genotype-phenotype" Correlations Observed in a Large Cohort of Patients With Hereditary Retinal Dystrophies - GEPHIRD
Acronym: GEPHIRD
Status: Terminated | Type: Observational
Why Stopped: Insufficient enrollment
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: EBA_2017_21
Record Dates: First submitted 2018-08-01; First posted 2018-09-07 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Retinal Dystrophies
Keywords: hereditary retinal dystrophies
MeSH Terms: interventions — Visual Acuity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspicion of hereditary retinal dystrophy
  Interventions: Procedure: OCT-A; Procedure: Visual acuity (ETDRS)

INTERVENTIONS:
Procedure: OCT-A — Optical coherence tomography angiography (OCT-A)
Procedure: Visual acuity (ETDRS) — Visual acuity tested with ETDRS score (Early Treatment Diabetic Retinopathy Study)

SUMMARY:
This study will carry out a detailed descriptive analysis of a large population of patients with hereditary retinal dystrophies (HRD): clinical, paraclinical and genetic data.

The information drawn from these analyzes will provide a better understanding of the pathophysiology of these rare diseases and this may ultimately impact the medical management of patients (targeted therapy).

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for suspicion of hereditary retinal dystrophy
* Benefiting as part of the care of a genetic analysis

Exclusion Criteria:

- Patient under a measure of legal protection

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized for suspicion of hereditary retinal distrophy
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Description of the phenotypic characteristics of patients with hereditary retinal dystrophies. | Baseline
  Phenotypic diagnosis of the type of retinal dystrophy based on all the examinations performed as part of the usual care and examinations added by the research (OCT-Angiography - Optical coherence tomography, and visual acuity with ETDRS scale : Early Treatment Diabetic Retinal Study, ETDRS).
Description of the genotypic characteristics of patients with hereditary retinal dystrophies. | Baseline
  Determination of the genetic mutations responsible for retinal dystrophy in order to confirm the phenotypic diagnosis and identify correlation between the phenotypic and genotypic characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Elise BOULANGER SCEMAMA, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation ophtalmologique Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided